CLINICAL TRIAL: NCT06378775
Title: Robotically-assisted Minimally-invasive Direct Coronary Artery Bypass With Stenting, Randomized Against Coronary Artery Bypass Graft Surgery: a Pilot Trial
Brief Title: Robotically-assisted Minimally-invasive Direct Coronary Artery Bypass With Stenting, Randomized Against Coronary Artery Bypass Graft Surgery
Acronym: ROBOT RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-03334
Record Dates: First submitted 2024-03-12; First posted 2024-04-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Multivessel Coronary Artery Disease
Keywords: CABG; Hybrid Coronary Revascularization; Robotically-assisted minimally-invasive direct coronary artery bypass; RA-MIDCAB
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Coronary Revascularization (Experimental): 2 Step revascularization: Robotically-assisted minimally-invasive direct coronary artery bypass (RA-MIDCAB) followed by Percutaneous Coronary Intervention (PCI)
  Interventions: Procedure: Robotically-assisted minimally-invasive direct coronary artery bypass; Procedure: Percutaneous Coronary Intervention
- Coronary Artery Bypass Grafting (CABG) (Active Comparator): Coronary Artery Bypass Grafting
  Interventions: Procedure: Coronary Artery Bypass Graft

INTERVENTIONS:
Procedure: Coronary Artery Bypass Graft — Coronary Artery Bypass Graft
  Other Names: CABG
  Arms: Coronary Artery Bypass Grafting (CABG)
Procedure: Robotically-assisted minimally-invasive direct coronary artery bypass — Robotically-assisted minimally-invasive direct coronary artery bypass
  Other Names: RA-MIDCAB
  Arms: Hybrid Coronary Revascularization
Procedure: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention
  Other Names: PCI
  Arms: Hybrid Coronary Revascularization

SUMMARY:
The study objective is to compare standard CABG to a hybrid revascularization strategy (RA-MIDCAB + PCI) in patients who have multi-vessel CAD and an indication for surgery, but who have a slightly higher risk of post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Multi-vessel CAD with an indication for revascularization,
2. Presence of at least 1 risk factor for increased risk of post-operative death or major complication,

   * Any patient Age > 80, OR
   * Any patient with eGFR (Glomerular Filtration Rate) < 50, OR
   * Any patient with LVEF < 40%, OR
   * Any patient deemed to be "frail" by consulting surgeon. OR
   * Patients > 75 years of age with at least one of the following:

     * Ejection fraction < 50%
     * History of prior CVA (Cerebral Vascular Accident)
3. Coronary artery anatomy appropriate for a robotically-assisted MIDCAB or regular CABG, vessels other than the left anterior descending with lesions amenable to either CABG or PCI.

Exclusion criteria

1. Significant left main coronary artery disease,
2. Ejection fraction < 30%,
3. Patients with GFR < 30,
4. Patients unable to take dual anti-platelet agents due to high bleeding risk,
5. Patients requiring emergent surgery, including patients with hemodynamic instability,
6. Patients with anatomy not suitable for a robotically-assisted approach (by CT chest).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative Length of Stay | From end of surgery (Skin time) to hospital discharge time, assessed up to 30 days
  Number of days from end of surgery to hospital discharge

SECONDARY OUTCOMES:
Conversion to sternotomy / CABG | From beginning of surgery time to end of surgery time (skin to skin)
  Rate of intraoperative conversion from RA-MIDCAB to sternotomy CABG (%)

OTHER OUTCOMES:
Intubation duration | From end of surgery time to extubation time
  Time to extubation post surgery measured in hours
ICU length of stay | From end of surgery time to ICU discharge time, assessed up to 10 days
  Time spent in ICU post-surgery measured in hours

IPD SHARING:
Plan to Share IPD: Undecided